CLINICAL TRIAL: NCT06114823
Title: Randomized Control Trial Comparing the Outcome of a Modified Mini-incision Approach Versus the Conventional Approach for Carpal Tunnel Release
Brief Title: Comparing a Modified Mini-incision Approach Versus the Conventional Approach for Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa, consultant and lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2345
Record Dates: First submitted 2023-10-20; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Carpal Tunnel Syndrome; Incision
MeSH Terms: conditions — Carpal Tunnel Syndrome; Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini incision group (Active Comparator): Patients were subjected to a longitudinal mini-incision started just above the proximal flexor wrist crease and then extended for 1.5 - 2 cm in a proximal direction.
  Interventions: Procedure: carpal tunnel release mini-incision; Procedure: carpal tunnel release conventional incision
- conventional group (Active Comparator): Patients were subjected a longitudinal incision which was created between the thenar and hypothenar eminences along the longitudinal axis of the ring finger. Then, it was extended to the proximal flexor wrist crease.
  Interventions: Procedure: carpal tunnel release mini-incision; Procedure: carpal tunnel release conventional incision

INTERVENTIONS:
Procedure: carpal tunnel release mini-incision — Patients were subjected to a longitudinal mini-incision started just above the proximal flexor wrist crease and then extended for 1.5 - 2 cm in a proximal direction
Procedure: carpal tunnel release conventional incision — Patients were subjected a longitudinal incision which was created between the thenar and hypothenar eminences along the longitudinal axis of the ring finger. Then, it was extended to the proximal flexor wrist crease.

SUMMARY:
Carpal tunnel syndrome (CTS) is the commonest nerve compression syndrome in the upper limbs, and carpal tunnel decompression is one of the most prevalent upper limb surgical interventions. Surgeries for CTS may be more effective compared to conservative measures in reducing symptoms and improving hand function, particularly in patients with severe CTS.

The etiology of CTS is multifactorial and includes occupational and personal factors. Physical workload factors play an important role in CTS but the role of some personal factors is less clear. Obesity is a well-documented risk factor for CTS. Hypothyroidism, diabetes mellitus, rheumatoid arthritis and osteoarthritis are possible risk factors for CTS. Finally, the role of smoking in CTS is uncertain.

Traditional approach makes use of a longitudinal skin incision from the palm toward the wrist and across the transverse carpal ligament. Though this approach offers excellent visualization, reliable release of the full retinaculum, and ability to identify anatomic variations, it is associated with some intractable complications, including wound pain, scar tenderness, flexor tendon entrapment and thenar as well as hypothenar (pillar) pain, which are difficult to recovery.

The attempt to perform CTR without extra complications leads to the development of different techniques and several mini-incision approaches.

These techniques help to reduce incisional discomfort after surgery, but it can lead to frequent incidence of blood vessel injury or incomplete release. The mini-incision approaches have the advantage of leaving a smaller scar, less scar pain, and lower grade of pillar pain. Though several methods have been proposed, there were still some disadvantages in them. Though CTR can be safely accomplished by them, incomplete release still occurred in several cases for some reasons.

After intensive research in the current literature, there is a paucity of studies evaluating the efficacy and safety of mini-incision approaches in achieving CTR in Egyptian patients. That is why we conducted the present study to present our experience with the modified mini-incision technique and compare its outcomes to the conventional open approach.

DETAILED DESCRIPTION:
All selected cases with primary CTS will be submitted to:

I) Preoperative evaluation:

A- Careful history taking: Brief history based on the characteristics of pain, sensory disturbances including numbness, tingling, and/or weakness involving the median nerve distribution. Patients were additionally inquired about their functional status, normal activities, ability to work, family history of diabetes and the use of medications.

B- The visual analogue scale (VAS) (0= no pain to 10= worst possible pain), will be used to assess the severity of diabetic neuropathic pain.

C- Neurosensory examination mainly included percussion over a distribution of the affected peripheral nerve (Tinel sign) and two-point discrimination (2-PD) using the Disk-Criminator.

D- Nerve conduction velocity (NCV).

II) Surgical Technique:

All patients are positioned on the operating table in supine position and anesthetized with local anaesthesia.

A) For the conventional approach: a palmar longitudinal incision began at the axis of the ring finger, passed between the thenar and hypothenar eminences, and continued proximally to the proximal flexor crease of the wrist. After exposing the underlying transverse carpal ligament, its ulnar side was cut longitudinally. The median nerve was identified and protected, and then the wound was closed in routine manner.

B) For the new mini-incision approach: a special metal guide with a groove at the center is used. The incision is started above the proximal flexor crease of the wrist and is advanced proximally for 1.5-2.0 cm. After opening the superficial fascia, blunt dissection with a mosquito clamp is performed till the median nerve appears and the guide is inserted into the carpal tunnel, then a scissor is inserted along the groove in the guide and the transverse carpal ligament is cut proximally and distally.

III) Postoperative follow up:

The follow-up was conducted mainly on an outpatient basis comparing the postoperative outcome in both groups as regard improvement of symptoms, postoperative complications, scar effect and recurrence of symptoms. Patients will be followed up at 2 weeks, 1 month, 3 months, and 6 months post decompression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary CTS attending Mansoura university hospitals with EMG-and NCS-proved median neuropathy at the wrist.
2. Failed conservative treatment.
3. Absence of any other hand pathology.
4. Positive Tinel sign presented at the site of nerve entrapment (the carpal tunnel at the wrist for the median nerve).
5. Signed informed consent.

Exclusion Criteria:

1. Presence of proximal radiculopathy.
2. Previous history of cervical spondylosis.
3. Inflammatory joint disease and gout.
4. Presence of combined nerve compression.
5. Having a previous hand or upper extremity surgery.
6. Patients with incomplete follow-up data were also excluded from this study.
7. Psychiatric disease or any other condition that is at risk of being inﬂuenced by the study or that might have affected completion of the study.
8. Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
improvement in carpal tunnel syndrome associated pain | 6 months postoperative
  According to visual analogue scale for pain which consists of 10 items , 0 for no pain and 10 for the maximum pain.

SECONDARY OUTCOMES:
pillar pain | 1,3&6 months postoperative
  According to visual analogue scale for pain which consists of 10 items , 0 for no pain or good outcome and 10 for the maximum pain or bad outcome.
recurrence of neuropathic symptoms | it will be evaluated till 6 months postoperative
  According to visual analogue scale for pain which consists of 10 items , 0 for no pain or good outcome and 10 for the maximum pain or bad outcome.
operative time | from start till the end of the operation
  From skin incision which is the start of the surgery ,till the end of the procedure
scar effect | from surgery till 3,6 months postoperative
  this item will measure the patients satisfaction for the skin scar as a cosmetic outcome, using the SCAR-Q scale which has 3 independently functioning scales that measure scar appearance, scar symptoms and its psychosocial impact.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed mahmoud, MD, Principal Investigator — Mansoura faculty of Medicine
Locations (1):
- Fuclty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No